CLINICAL TRIAL: NCT06293599
Title: Effect of Scapular Stabilization Exercises Versus Virtual Reality Exercises in Basketball Players With Scapular Dyskinesia
Acronym: SD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nabil Mahmoud Ismail Abdel-Aal, Principal investigator Nabil mahmoud ismail, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003131
Record Dates: First submitted 2024-01-31; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Scapular Dyskinesis
Keywords: scapular stabilization; virtual reality; scapular dyskinesia
MeSH Terms: interventions — Exergaming

STUDY DESIGN:
Intervention Model Description: scapular stabilization and virtual reality exercise
Who Masked: Investigator, Outcomes Assessor
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- scapular stabilization exercise (Experimental): thirty patients with scapular dyskinesia will receive scapular stabilization exercise and regular routine three times a week for eight weeks
  Interventions: Other: scapular stabilization exercises; Other: regular routine exercises
- virtual reality exercise (Experimental): thirty patients with scapular dyskinesia will receive virtual reality exercise and regular routine three times a week for eight weeks
  Interventions: Other: virtual reality exercises; Other: regular routine exercises
- Regular routine exercise (Active Comparator): thirty patients with scapular dyskinesia will receive regular routine exercises three times a week for eight weeks
  Interventions: Other: regular routine exercises

INTERVENTIONS:
Other: scapular stabilization exercises — the patients will receive scapular stabilization exercises in the form of scapular orientation exercises,Forward/Backward Bear Crawls,Lateral Bear Crawls and assisted stretch for pectoralis minor
  Arms: scapular stabilization exercise
Other: virtual reality exercises — The exercises described were done in a consistent manner, emphasizing low intensity, and using lightweight dumbbells (range, 3 to 30 pounds). The weight of the dumbbell was individually selected by the subject for each exercise.
  1. elevation of the arm in the sagittal plane (shoulder flexion
  2. elevation of the arm in the scapular plane with humeral external rotation (shoulder scaption
  3. elevation of the arm in the coronal plane (shoulder abduction)
  4. rowing
  5. horizontal shoulder abduction
  6. horizontal abduction with humeral external rotation
  7. push-up with hands apart
  8. push-up with a plus-normal push-up adding maximum shoulder and scapular protraction with elbows fully extended
  9. dumbbell bench press
  10. dumbbell military press
  11. shoulder shrug
  12. deceleration exercise-simulating the pitching followthrough
  13. shoulder extension prone
  14. shoulder internal rotation
  15. shoulder external rotation
  16. press-up
  Arms: virtual reality exercise
Other: regular routine exercises — the patients will receive routine exercises in the form of Sleeper Stretch: Posterior Capsular Stretch, Push up, Wall slides, Kettlebell High Pull,

SUMMARY:
this study will be conducted to compare virtual reality and scapular stabilizing exercise among basketball player with scapular dyskinesia on scapular muscle performance, rounded shoulder, pain intensity , disability and hand grip strength

DETAILED DESCRIPTION:
Scapular dyskinesia (SD) is an alteration in the normal position or motion of the scapula during coupled scapulohumeral movements. It is lack of control of static or dynamic positioning of the scapula relative to the thorax. It affects from 64% to 100% of patients with shoulder lesions. Scapular dyskinesia is a major etiological factor in overhead athletes' shoulder problems. Virtual Reality (VR) it allows individuals to interact and train with or within interesting and relatively realistic three-dimensional(3D) environments. VR and its simulated environments are well accepted in entertainment and computer game applications. However, what is not as well recognized is that VR offers the opportunity for intensive repetition of meaningful task-related activities necessary for effective rehabilitation. The scapular stabilization exercise in rehabilitation aims to Restore shoulder function; these exercises are a combination of scapular stabilization exercises, rotator cuff strengthening exercises, range of motion (ROM), proprioceptive neuromuscular facilitation (PNF), and stretching exercises. Physiotherapy is the mainstay management for several musculoskeletal disorders. sixty basketball athletes with dyskinesea will be assigned randomly to three equal groups; the first will receive Virtual reality exercise and routine exercise, and the second group will receive Stabilization exercise and routine exercise. and finally, the third group will receive routine exercise only for eight weeks

ELIGIBILITY:
Inclusion Criteria:

* ninety basketball players of both genders.
* Subjects with age between 20 and 25 years old.
* Subjects with Body Mass Index (BMI) ranging from 18 to 25 kg/m².

Exclusion Criteria:

* An injury within the four weeks before testing.
* Upper extremity fractures.
* Bilateral repetitive strain injuries
* Osteoarthritis on hand

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-03-05 (Estimated); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
agonist antagonist ratio | up to eight weeks
  isokinetic Biodex 3 dynamometer will be used to assess agonist antagonist ratio

SECONDARY OUTCOMES:
Hand grip strength | up to eight weeks
  Jamar handheld dynamometer will be used to assess hand grip strength
rounded shoulder posture | up to eight weeks
  Patient is supine with the arms at the sides, elbows extended, palms upward, knees bent and lower back flat on the table. The examiner stands at the head of the table and use tape measurements to measure the distance between the acromion of the shoulder joint and the table surface three times. The numbers were averaged and used for analysis. Increased distance signifies higher rounded shoulder posture severity
pain intensity level | up to eight weeks
  Visual Analogue Scale (VAS) will be used to assess pain by Using a ruler, the score is determined by measuring the distance on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-10. A higher score indicates greater pain intensity.
The disabilities of the arm, shoulder and hand | up to eight weeks
  The disabilities of the arm, shoulder and hand (DASH) questionnaire will be used to assess the disability in arm, shoulder and hand. The DASH consists mainly of a 30- item disability/symptom scale. The possible score ranges from 0 to 100 points. 0 points represent a complete, unrestricted function of the upper extremities, while 100 points represent the greatest possible functional impairment.
peak force | up to eight weeks
  isokinetic Biodex 3 dynamometer will be used to assess peak force
total work | up to eight weeks
  isokinetic Biodex 3 dynamometer will be used to assess total work
work fatigue | up to eight weeks
  isokinetic Biodex 3 dynamometer will be used to assess work fatigue
average power | up to eight weeks
  isokinetic Biodex 3 dynamometer will be used to assess average power